CLINICAL TRIAL: NCT05469334
Title: DeStress for Health: Partnering With Granville and Vance Counties to Reduce Stress and Cancer Risk
Brief Title: DeStress for Health: Partnering With Granville and Vance Counties to Reduce Stress and Cancer Risk (Part 2)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00100183_1
Record Dates: First submitted 2022-07-19; First posted 2022-07-21 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Stress Reduction
Keywords: Stress Reduction; Rural; North Carolina; Health Behaviors
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: DeStress for Health Program Participants (Experimental): Rural residents 18 years and older of Granville and Vance counties (n=40) will be recruited to participate.
  Interventions: Behavioral: DeStress for Health Program Participants

INTERVENTIONS:
Behavioral: DeStress for Health Program Participants — Behavioral: DeStress for Health Program The program will consist of 4 in person sessions that are based on empirically supported Positive Psychosocial Well-Being PPWB components including Optimism, Mindfulness, Positive Reprisal as well as Strengths-based Cognitive Behavioral Therapy (SBCBT) to improve behavioral self-regulation towards health-related goals, with an additional class five as a check in that will be used for survey completion. Research staff will conduct face-to-face surveys with participants at baseline and at end of program. Finally, we will conduct a phone-based survey 30 days after program completion to assess sustainability of intervention effects.

SUMMARY:
The purpose of this research study is to determine whether a positive psychology intervention paired with a health behavior intervention is successful in decreasing perceived stress and increasing positive affect in residents of Vance and Granville County.The program will consist of 4 in person / zoom sessions that are based on empirically supported PPWB components including Optimism, Gratitude, Mindfulness and Positive Savoring to improve behavioral self-regulation towards health-related goals with an additional class five as a check in that will be used for survey completion. Specifically, principal investigator will provide participants with instruction on positive psychology exercises that can do on their own and counseling around increased fruit and vegetable intake, physical activity and smoking cessation. Participants will then be asked to create a SMART goal to work on each week of the program for one of the behaviors. Research staff will conduct surveys with participants at baseline and at end of program. Feasibility and acceptability measures of the intervention will be collected at the end of the program. Research team will also collect informal feedback from participants at the end of each of the class sessions. Classes will be delivered in person and broadcasted via zoom via a password protected zoom link. Participant who choose to remain remote and participate via Zoom will be mailed binders of study materials with information on who to call if participants have questions. Participants who attend live events will receive their materials in person. Pre- and post-intervention surveys will be sent to participants via email. This is Part 2 of study (NCT03776890)

ELIGIBILITY:
Inclusion Criteria:

* Live in Granville or Vance Counties;
* >18 years old;
* Interested in participating a stress reduction study
* Speak English

Exclusion Criteria:

* Does Not Live in Granville or Vance Counties
* Under 18 years of age
* Not interested in participating in a stress reduction study
* does not speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
Number of Participants Recruited in a 6-Month Time-frame | 6 months
  Measured via subject enrollment log
Percentage of Participants That Stay in Study for Duration | 2 months
  Measured via subject enrollment log
Percentage of Participants That Attend All Intervention Sessions | 2 months
  Measured via subject enrollment log
Percent of Participants Rating Intervention as Useful | 2 months
  Measured on a scale from 1-5 with 1 being "Not Useful at All" and 5 being "Extremely Useful".
Percent of Participants Recommending Intervention to Friend | 2 months
  Measured on a scale from 1-5 with 1 being "Not at All" and 5 being "Extremely".

SECONDARY OUTCOMES:
Change in Stress Self Regulation As Measured By a Survey | 2 months
  qualitative scale I agree a lot I agree a little I neither agree nor disagree I disagree a little I disagree a lot
Change in Positive Emotion As Measured by a Survey | 2 months
  qualitative scale I agree a lot I agree a little I neither agree nor disagree I disagree a little I disagree a lot
Change in Behavioral Self Regulation As Measured by a Survey | 2 months
  qualitative scale I agree a lot I agree a little I neither agree nor disagree I disagree a little I disagree a lot

CONTACTS AND LOCATIONS:
Overall Officials: Devon Noonan, Ph.D, Principal Investigator — Duke School of Nursing
Locations (1):
- Granville Vance Public Health Department, Oxford, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No